CLINICAL TRIAL: NCT05250752
Title: Reduction of Peritoneal Glucose Uptake With Use of SGLT2 in Humans Undergoing Peritoneal Dialysis Treatment. A Proof of Concept Phase 2a Clinical Trial.
Brief Title: Reduction of Peritoneal Glucose Uptake With Use of SGLT2 in Humans Undergoing Peritoneal Dialysis Treatment
Acronym: PRESERVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOL-MED-01-2021
Record Dates: First submitted 2022-01-13; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-11

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis Complication
Keywords: SGLT2-inhibition; dapagliflozin
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Cross-over. Off-On-Off treatment. Dose response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- On treatment (Other): Assigned to oral treatment with dapagliflozin 10 mg for three consecutive days.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Primary end-points are measure before (day 0), on treatment (day 1 and day 3) and after treatment (day 21)

SUMMARY:
End stage renal disease is annually diagnosed in about one thousand patients in Denmark, and one of the treatment modalities in renal replacement therapy is peritoneal dialysis with about 25 % of patients assigned to this treatment (Hommel2010). Peritoneal dialysis is based on the principle of filtering waste products to peritoneal fluid and by exchange of peritoneal fluid eliminate waste products from the body.

In peritoneal dialysis commonly used fluids contain glucose. Exposure to high glucose levels in peritoneal fluid during peritoneal dialysis has several side effects. Primarily, as glucose passes over and into the peritoneal membrane it causes local inflammation which leads to fibrosis over time (Zhou2016). Fibrosis limits the capacity of the exchange of water and waste products over the peritoneal membrane. The decrease of peritoneal exchange capacity is most commonly the reason for termination of peritoneal dialysis.

SGLT2-channels are identified in peritoneal mesothelial cells of rats (Debray-Carcia 2016), and most recently also in humans (Shentu2021). An in vitro model of human peritoneal mesothelial cells incubated with the SGLT2-inhibitor (empagliflozin) has shown significantly decrease in glucose uptake (Zhou2019). Exposure to intraperitoneal empagliflozin in rats, reduced the uptake of glucose over the peritoneal membrane significantly by 78 % and the ultrafiltration was increased (Zhou2019).

Currently, to our knowledge, no clinical trials have been conducted in humans attending peritoneal dialysis with the aim of investigating either the effect or safety of SGLT2i, as it is indeed the first of its kind, with the aim of including participants in peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age above 18 years of age
3. In stable peritoneal dialysis for more than 14 days.

Exclusion Criteria:

1. In treatment with SGLT2i currently or within the last 90 days.
2. Treatment for peritoneal infection within the last 30 days.
3. Any hospitalization within the last 30 days.
4. Anaphylaxis to the IMP.
5. Impaired lever function with ALAT above normal range within the last 6 month.
6. Sever efflux problems during peritoneal dialysis for the last 14 days, judged by the investigator.
7. Non-menopausal defined as menstruation within the last 12 month without any other medical cause. Only applicable for female participants.
8. Substance abuse, judged by the investigator.
9. Incapable to follow study protocol, judged by the investigator.
10. Previously included in this clinical trial and exposed to the IMP.
11. Included in another clinical trial with exposure to any IMP within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-02-27 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Peritoneal glucose uptake (mg/ dL) | Day 0 (baseline), Day 3 (max dose of treatment)
  Glucose level in peritoneal fluid during a four hour standardized peritoneal dialysis. Change in total glucose uptake before and after treatment (treatment periode of three days)

SECONDARY OUTCOMES:
Fluid volume (ml) | Measured at end of each peritoneal dialysis. Peritoneal dialysis done af Day 0, Day 1 (first day of treatment) and day 3 (max dose of treatment)
  Fluid volume ultra-filtrated during peritoneal dialysis.
Plasma glucose level (mg/ dL) | Measured at end of each peritoneal dialysis. Peritoneal dialysis done af Day 0, Day 1 (first day of treatment) and day 3 (max dose of treatment).
  Glucose levels in blood and peritoneal-fluid during peritoneal dialysis. Comparaison of maximal plasma level.
Pharmacokinetics (nmol) | Samples for biobank - samples drawn at end of each peritoneal dialysis. Peritoneal dialysis done af Day 0, Day 1 (first day of treatment) and day 3 (max dose of treatment). Samples are drawn every 30 minuttes during each peritoneal dialysis.
  Dapagliflozin and its metabolites levels in blood and peritoneal-fluid
Adverse events (events) | At day 1 (first day of treatment), day 3 (max dose of treatment) and day 30 (four weeks after treatment)
  Safety in terms of AE and/or SAE

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindhardt, MD, PhD, Principal Investigator — Copenhagen University Hospital - Holbaek
Locations (1):
- University Hospital Copenhagen - Holbaek, Holbæk, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data material used in this study are available from the corresponding author on reasonable request which will not conflict with the anonymity and confidentiality of the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Depended on the request - Days to weeks
Access Criteria: Not conflict with the anonymity and confidentiality of the data and a signed contract for data sharing.